CLINICAL TRIAL: NCT02332980
Title: A Phase II Study of Anti-PD-1 Antibody (MK-3475) in Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL) and Other Low Grade B Cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Pembrolizumab Alone or With Idelalisib or Ibrutinib in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Other Low-Grade B-Cell Non-Hodgkin Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1485; NCI-2014-02561 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1485 (Other: Mayo Clinic in Rochester); P50CA097274 (NIH); 14-005666 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Results first posted 2023-03-21 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Lymphoplasmacytic Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Nodal Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Recurrent Splenic Marginal Zone Lymphoma; Recurrent Waldenstrom Macroglobulinemia; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Refractory Follicular Lymphoma; Refractory Lymphoplasmacytic Lymphoma; Refractory Nodal Marginal Zone Lymphoma; Refractory Small Lymphocytic Lymphoma; Refractory Splenic Marginal Zone Lymphoma; Refractory Waldenstrom Macroglobulinemia; Richter Syndrome; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Waldenstrom Macroglobulinemia | interventions — ibrutinib; idelalisib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pembrolizumab, idelalisib, or ibrutinib) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients receiving benefit may continue to receive treatment for an additional 12 months at the discretion of the investigator. Patients with CLL or CLL with Richter's transformation experiencing stable disease without partial remission or progressive disease at 3 months of treatment with pembrolizumab proceed to the treatment continuation phase.
  CONTINUATION PHASE: Patients receive pembrolizumab IV over 30 minutes on day 1. Patients also receive idelalisib PO BID on days 1-21 OR ibrutinib PO QD on days 1-21. Treatment repeats every 21 days for up to 12 or 24 months in the absence of disease progression or unacceptable toxicity. Patients receiving benefit may continue to receive treatment for an additional 12 months at the discretion of the investigator.
  Interventions: Drug: Ibrutinib; Drug: Idelalisib; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Idelalisib — Given PO
  Other Names: CAL-101; GS 1101; GS-1101; Phosphoinositide-3 Kinase Delta Inhibitor CAL-101; Zydelig
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab alone or with idelalisib or ibrutinib works in treating patients with chronic lymphocytic leukemia or other low-grade B-cell non-Hodgkin lymphomas that have returned after a period of improvement (relapsed) or have not responded to treatment (refractory). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Idelalisib and ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab alone or with idelalisib or ibrutinib may be an effective treatment in patients with chronic lymphocytic leukemia or other low-grade B-cell non-Hodgkin lymphomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Test the efficacy (overall response rate) of single-agent MK-3475 (pembrolizumab) in relapsed chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) (Arm A) other low grade B-cell non-Hodgkin lymphoma (B-NHL), and CLL with Richter's transformation (Arm C).

SECONDARY OBJECTIVES:

I. Test the safety of single-agent MK-3475 in relapsed CLL/SLL (Arm A), other low grade B-NHL (Arm B), and CLL with Richter's transformation (Arm C).

II. Test the overall survival, progression free survival, treatment free survival, duration of response and time to next therapy of single-agent MK-3475 in relapsed CLL/SLL (Arm A), other low grade B-NHL (Arm B), and CLL with Richter's transformation (Arm C).

III. Test the complete response rate of single MK-3475 in relapsed CLL/SLL (Arm A), other low grade B-NHL (Arm B), and CLL with Richter's transformation (Arm C).

IV. Test the safety of MK-3475 in combination with the signal inhibitor (either idelalisib or ibrutinib) in relapsed CLL/SLL (Arm A) and CLL with Richter's transformation (Arm C).

V. Test the progression-free survival, treatment-free survival, duration of response and time to next therapy, as well as overall survival of MK-3475 in combination with the signal inhibitor (either idelalisib or ibrutinib) in relapsed CLL/SLL (Arm A) and CLL with Richter's transformation (Arm C).

VI. Test the overall and complete response rates of MK-3475 in combination with the signal inhibitor (either idelalisib or ibrutinib) in relapsed CLL/SLL (Arm A) and CLL with Richter's transformation (Arm C).

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess the potential association between programmed cell death ligand 1 (PD-L1)/programmed cell death 1 (PD-1)/PD-L2 expression on tumor and T cells and/or PD-L1 soluble levels in plasma with clinical efficacy of PD-1 blockade.

II. To investigate the effects of MK-3475 on selected markers of immune modulation and immune profiles in peripheral blood and tumor samples.

III. Examine T-cell immune synapse function and expression/location of co-stimulatory and co-inhibitory molecules (including effector molecules) as potential biomarkers to response for anti-PD-1 immune checkpoint blockade immunotherapy.

OUTLINE:

ALL PATIENTS (ARMS A, B, and C): Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients receiving benefit may continue to receive treatment for an additional 12 months at the discretion of the investigator. Patients with CLL or CLL with Richter's transformation experiencing stable disease without partial remission or progressive disease at 3 months of treatment with pembrolizumab proceed to the treatment continuation phase.

CONTINUATION PHASE (ARMS A and C): Patients receive pembrolizumab IV over 30 minutes on day 1. Patients also receive idelalisib orally (PO) twice daily (BID) on days 1-21 OR ibrutinib PO once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 12 or 24 months in the absence of disease progression or unacceptable toxicity. Patients receiving benefit may continue to receive treatment for an additional 12 months at the discretion of the investigator.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* CLL/SLL PATIENTS (ARM A) ONLY
* Diagnosis of CLL according to the National Cancer Institute (NCI) criteria or SLL according to the World Health Organization (WHO) criteria; this includes previous documentation of:

  * Biopsy-proven small lymphocytic lymphoma or
  * Diagnosis of CLL according to NCI working group criteria as evidenced by all of the following:

    * Peripheral blood B cell count of > 5 x 10^9/L consisting of small to moderate size lymphocytes
    * Immunophenotyping consistent with CLL defined as:

      * The predominant population of lymphocytes share both B-cell antigens (cluster of differentiation [CD]19, CD20 [typically dim expression] or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc.)
      * Clonality as evidenced by kappa or lambda light chain expression (typically dim immunoglobulin expression) or other genetic method (e.g. immunoglobulin heavy chain variable [IGHV] analysis)
      * NOTE: splenomegaly, hepatomegaly, or lymphadenopathy are not required for the diagnosis of CLL
    * Before diagnosing CLL or SLL, mantle cell lymphoma must be excluded by demonstrating a negative fluorescent in situ hybridization (FISH) analysis for t(11;14) (immunoglobulin H [IgH]/cyclin D1 [CCND1]) on peripheral blood or tissue biopsy or negative immunohistochemical stains for cyclin D1 on involved tissue biopsy
* Patients must be previously treated with at least one prior line of therapy; EXCEPTION: CLL patients with Richter's transformation or Hodgkin transformation do not need prior therapy to enroll

  * NOTE:

    * Prior chemotherapy or biologic novel therapy or anti-cancer monoclonal antibody based therapy for treatment of CLL will be considered prior therapy; nutraceutical treatments with no established benefit in CLL (such as epigallocatechin gallate or EGCG, found in green tea or other herbal treatments) will not be considered "prior treatment"
    * Prior oral corticosteroid therapy for an indication other than CLL will not be considered "prior treatment"
    * Previous use of corticosteroids in the combination with other therapy for treatment of autoimmune complications of CLL does constitute prior therapy for CLL
* CLL/SLL patients must have progressive disease with any one of the following characteristics based on standard criteria for treatment as defined by the NCI-Working Group (WG) 1996

  * Symptomatic CLL characterized by any one of the following:

    * Weight loss >= 10% within the previous 6 months
    * Extreme fatigue attributed to CLL
    * Fevers >= 100.5 degree Fahrenheit (F) for 2 weeks without evidence of infection
    * Drenching night sweats without evidence of infection
  * Evidence of progressive bone marrow failure with hemoglobin =< 11 g/dL or platelet count =< 100 x 10^9/L
  * Symptomatic or progressive lymphadenopathy, splenomegaly, or hepatomegaly
  * Note: marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease are not sufficient for protocol therapy OR biopsy proven Richter's transformation or Hodgkin transformation of the CLL; NOTE: both untreated and previously treated patients in this category can be enrolled; they do not need to meet the progressive disease criteria in first bullet as long as measurable disease can be detected by positron emission tomography (PET)/computed tomography (CT) or CT (>= 1.5 cm in diameter)
* LOW GRADE B-NHL PATIENTS ONLY
* Histologically confirmed relapsed (response to last treatment >= 6 months duration) or refractory (no response to last treatment or response duration < 6 months) indolent/low grade B cell NHL; NOTE: if patient has received previous anti-PD-1 or anti-PDL-1 consult with study chair

  * Follicular lymphoma, grades 1, 2 and 3
  * Extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue (MALT) type
  * Splenic and nodal marginal zone lymphoma
  * Lymphoplasmacytic lymphoma including Waldenstrom macroglobulinemia
* Measurable disease (at least 1 lesion of >= 1.5 cm in diameter) as detected by CT or the CT images of the PET/CT; NOTE: patients with Waldenstrom macroglobulinemia are not required to have measurable disease by CT or PET/CT if monoclonal protein is detectable by serum protein electrophoresis and/or immunoglobulin M (IgM) level is at least 2 times upper limit of normal
* CLL WITH RICHTER's TRANSFORMATION (ARM C) ONLY
* CLL diagnosis confirmed as have biopsy-proven Richter's transformation; NOTE: both untreated and previously treated patients in this category can be enrolled as long as measurable disease can be detected by PET/CT or CT (>= 1.5 cm in diameter)
* ALL PATIENTS
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Creatinine =< 1.5 x upper limit of normal (ULN) OR creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (obtained =< 14 days prior to registration)
* Platelet count >= 25 x 10^9/L (obtained =< 14 days prior to registration)
* Absolute neutrophil count >= 0.5 x 10^9/L (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilbert's disease; if total bilirubin is > 1.5 x ULN, a direct bilirubin should be performed and must be =< upper limit of normal (obtained =< 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN (obtained =< 14 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

  * Note: During the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide bone marrow, tissue, and blood samples for correlative research purposes
* Must have failed or be unable to tolerate or refused other available Food and Drug Administration (FDA) approved effective therapies; NOTE: patients should not have other treatment options considered curative

Exclusion Criteria:

* Currently participating in or has participated in a study of an investigational agent or using an investigational device =< 28 days prior to registration
* Receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy =< 7 days prior to registration; EXCEPTIONS:

  * Low doses of steroids (=< 20 mg of prednisone or equivalent dose of other steroid/day)
  * Previous use of corticosteroids is allowed
  * After initiation of MK-3475 therapy, steroid can be used for management of potential immune mediated adverse events (AE) for less than 8 weeks of therapy
  * Topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption) are permitted
* Prior anti-cancer monoclonal antibody =< 28 days prior to registration or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Prior chemotherapy or radiation therapy =< 14 days prior to registration or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Known additional malignancy that is progressing or requires active treatment; EXCEPTIONS (these following exceptions are permitted to enroll in this trial):

  * Basal cell carcinoma or squamous cell carcinoma or melanoma of the skin that has undergone or will undergo potentially curative therapy
  * In situ cervical cancer that has undergone or will undergo potentially curative therapy
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease/syndrome difficult to control in the past; EXCEPTIONS:

  * Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule
  * Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study
  * Subjects with hypothyroidism stable on hormone replacement, diabetes or Sjogren's syndrome are permitted for the study
  * Patients who have a positive Coombs test but no evidence of hemolysis are permitted for participation
  * Patients with psoriasis not requiring systemic treatment are permitted for participation
  * Conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Evidence of interstitial lung disease or active, non-infectious pneumonitis
* Active infection requiring systemic therapy; NOTE: when the infection is controlled, patients are permitted for this study
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Known to be human immunodeficiency virus (HIV) positive
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected); NOTE: patients with active hepatitis B defined by hepatitis B surface antigen positivity or core antibody positivity in the presence of hepatitis B deoxyribonucleic acid (DNA) are not eligible for this study; patients with a positive hepatitis B core antibody but with negative hepatitis B DNA may participate, but must have hepatitis serologies and hepatitis B DNA monitored periodically by the treating physician

  * NOTE: intravenous immunoglobulin (IVIG) can cause a false positive hepatitis B serology; if patients receiving routine IVIG have core antibody or surface antigen positivity without evidence of active viremia (negative hepatitis B DNA) they may still participate in the study, but should have hepatitis serologies and hepatitis B DNA monitored periodically by the treating physician
* Received a live vaccine =< 30 days prior to registration
* New York Heart Association classification III or IV cardiovascular disease or recent myocardial infarction or unstable angina pectoris or cardiac arrhythmia (< 30 days)
* Active central nervous system (CNS) lymphoma or cerebrospinal fluid involvement with malignant lymphoma cells that requires therapy
* Has a clinically significant coagulopathy per investigator's assessment
* Has received an allogeneic stem cell transplant
* CLL ARMS (ARM A and ARM C) FOR COMBINATION THERAPY INCLUDING IBRUTINIB or IDELALISIB:
* Is chronically taking a strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A) inhibitor or inducer and cannot be switched to an alternative agent at least 7 days prior to idelalisib or ibrutinib initiation that in the opinion of investigator/treating physicians precludes utilization of either Ibrutinib or Idelalisib; caution is recommended for patients taking moderate inhibitors of CYP3A
* CLL ARMS (ARM A and ARM C) FOR COMBINATION THERAPY INCLUDING IDELALISIB ARM:
* Is chronically taking a sensitive CYP3A substrate or a CYP3A substrate with a narrow therapeutic index and cannot be switched to an alternative agent at least 7 days prior to study initiation that in the opinion of investigator/treating physicians precludes utilization of idelalisib
* A history of chronic diarrhea, colitis, or intestinal perforation that in the opinion of the investigator precludes utilization of idelalisib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Ding, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Ding W, LaPlant BR, Call TG, Parikh SA, Leis JF, He R, Shanafelt TD, Sinha S, Le-Rademacher J, Feldman AL, Habermann TM, Witzig TE, Wiseman GA, Lin Y, Asmus E, Nowakowski GS, Conte MJ, Bowen DA, Aitken CN, Van Dyke DL, Greipp PT, Liu X, Wu X, Zhang H, Secreto CR, Tian S, Braggio E, Wellik LE, Micallef I, Viswanatha DS, Yan H, Chanan-Khan AA, Kay NE, Dong H, Ansell SM. Pembrolizumab in patients with CLL and Richter transformation or with relapsed CLL. Blood. 2017 Jun 29;129(26):3419-3427. doi: 10.1182/blood-2017-02-765685. Epub 2017 Apr 19. PMID 28424162

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (CLL); Arm C (CLL With Richters): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients receiving benefit may continue to receive treatment for an additional 12 months at the discretion of the investigator. Patients on Arm A or Arm C experiencing stable disease without partial remission or progressive disease at 3 months of treatment with pembrolizumab proceed to the treatment continuation phase.
- Arm B (NHL): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients receiving benefit may continue to receive treatment for an additional 12 months at the discretion of the investigator.
Period: Initial Study Phase
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters)
Started | 25 | 23 | 17
Completed | 25 | 23 | 17
Not Completed | 0 | 0 | 0
Period: Continuation Phase
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters)
Started | 5 | 0 | 13
Completed | 5 | 0 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters) | Total
Number analyzed (Participants) | 25 | 23 | 17 | 65
Age, Continuous [Median (Full Range); unit: years] | 69 [46 to 81] | 67 [47 to 82] | 68 [57 to 83] | 69 [46 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 6 | 23
  Male | 17 | 14 | 11 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 20 | 15 | 57
  Unknown or Not Reported | 3 | 3 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 25 | 22 | 15 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieve a Confirmed Response
Description: Confirmed response is defined to be a partial response, nodular partial response, clinical complete response, confirmed response with incomplete blood count recovery or confirmed response (Arm A and B), or complete metabolic response, partial metabolic response, partial response, or confirmed response (Arm C). The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial confidence intervals for the true success proportion will be calculated.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: proportion of responders
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters)
Number analyzed (Participants) | 25 | 23 | 17
proportion of responders | 0.0800 [0.0098 to 0.2603] | 0 [0 to 0.1482] | 0 [0 to 0.1951]

2. Secondary Outcome: Progression-free Survival of Patients Treated in Single Agent Phase
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters)
Number analyzed (Participants) | 25 | 23 | 17
Months | 2.8 [1.4 to 4.6] | 4.2 [2.6 to 6.4] | 2.2 [0.7 to 2.8]

3. Secondary Outcome: Progression-free Survival of Patients Treated With Combination Therapy
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A (Continuation Phase); Arm C (Continuation Phase): CONTINUATION PHASE: Patients receive pembrolizumab IV over 30 minutes on day 1. Patients also receive idelalisib PO BID on days 1-21 OR ibrutinib PO QD on days 1-21. Treatment repeats every 21 days for up to 12 or 24 months in the absence of disease progression or unacceptable toxicity. Patients receiving benefit may continue to receive treatment for an additional 12 months at the discretion of the investigator.
Arm/Group | Arm A (Continuation Phase) | Arm C (Continuation Phase)
Number analyzed (Participants) | 5 | 13
Months | 7.6 [1.9 to NA] — Not enough events occurred to calculate upper limit | 5.4 [0.7 to 15.0]

4. Secondary Outcome: Treatment-free Survival of Patients Treated With Single-agent Pembrolizumab
Description: The distribution of treatment-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters)
Number analyzed (Participants) | 25 | 23 | 17
Months | 2.7 [2.1 to 3.2] | 4.6 [3.1 to 8.1] | 2.9 [0.8 to 3.4]

5. Secondary Outcome: Treatment-free Survival of Patients Treated With Combination Therapy
Description: The distribution of treatment-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Continuation Phase) | Arm C (Continuation Phase)
Number analyzed (Participants) | 5 | 13
Months | 7.7 [0.7 to NA] — Not enough events occurred to calculate upper limit | 3.2 [0.5 to 5.1]

6. Secondary Outcome: Time to Next Treatment for Patients Treated With Single-agent Pembrolizumab
Description: The distribution of time to next treatment will be estimated using the method of Kaplan-Meier.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters)
Number analyzed (Participants) | 25 | 23 | 17
Months | 3.0 [2.1 to 3.9] | 5.3 [3.4 to 10.1] | 3.0 [1.1 to 3.4]

7. Secondary Outcome: Time to Next Treatment for Patients on Combination Therapy
Description: The distribution of time to next treatment will be estimated using the method of Kaplan-Meier.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Continuation Phase) | Arm C (Continuation Phase)
Number analyzed (Participants) | 5 | 13
Months | 7.7 [0.7 to NA] — Not enough events occurred to calculate upper limit | 3.2 [0.5 to 5.1]

8. Secondary Outcome: Complete Response Rate
Description: Will be defined as complete response or incomplete blood count recovery. Estimated by the number of patients who achieve an incomplete blood count recovery or complete response divided by the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true complete response rate will be calculated in each arm.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters) | Arm A (Continuation Phase) | Arm C (Continuation Phase)
Number analyzed (Participants) | 25 | 23 | 17 | 5 | 13
proportion of participants | 0.0400 [0.0010 to 0.2035] | 0 [0 to 0.1482] | 0 [0 to 0.1951] | 0.4000 [0.0527 to 0.8534] | 0 [0 to 0.2471]

9. Secondary Outcome: Duration of Response
Description: The distribution of duration of response will be estimated using the method of Kaplan-Meier. Duration of response (DR) is defined for all evaluable patients who have achieved a PR, nPR, CCR, CRi, or CR (Arms A and B) or PMR, CMR, PR or CR (Arm C) as the date at which the patient's objective status is first noted to be a PR, nPR, CCR, CRi, or CR (Arms A and B) or PMR, CMR, PR or CR (Arm C) to the earliest date relapse is documented.
Time Frame: 5 years
Population: Only patients that achieved a response were used in this analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters) | Arm A (Continuation Phase) | Arm C (Continuation Phase)
Number analyzed (Participants) | 2 | 0 | 0 | 5 | 13
Months | 6.9 [2.6 to NA] — Not enough events occurred for upper limit calculation |  |  | 5.9 [2.6 to NA] — Not enough events occurred for upper limit calculation | NA [10.7 to NA] — Not enough events occurred for median or upper limit calculation

10. Secondary Outcome: Overall Survival
Description: The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters) | Arm A (Continuation Phase) | Arm C (Continuation Phase)
Number analyzed (Participants) | 25 | 23 | 17 | 5 | 13
Months | 10.6 [5.4 to 34.4] | 48.6 [13.0 to NA] — Not enough events to estimate upper confidence limit | 11.5 [4.1 to 17.6] | 11.7 [1.9 to NA] — Not enough events to estimate upper confidence limit | 13.3 [5.8 to NA] — Not enough events to estimate upper confidence limit

11. Secondary Outcome: Confirmed All Response Rate of Patients Treated With Combination Therapy
Description: Confirmed response rate will be estimated by the number of patients with an objective status of complete response, incomplete blood count recovery, nodular partial response, clinical complete response or partial response while on the combination therapy divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall response rate to the combination will be calculated. In addition, the responders on this study will be further examined in an exploratory manner to determine if there are any patterns in prognostic factors or disease characteristics, including whether the patient had a Richter's transformation or ibrutinib-resistant disease, for both single agent pembrolizumab and combination therapy responders.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Continuation Phase) | Arm C (Continuation Phase)
Number analyzed (Participants) | 5 | 13
proportion of participants | 0.6000 [0.1466 to 0.9473] | 0.1538 [0.0192 to 0.4545]

12. Secondary Outcome: Incidence of Adverse Events
Description: Will be measured per National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Adverse events will be evaluated for single-agent pembrolizumab in each arm and also for the combination of pembrolizumab and the signal inhibitor in Arm A and Arm C. This outcome is reported in the adverse events section of this report.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters) | Arm A (Continuation Phase) | Arm C (Continuation Phase)
Number analyzed (Participants) | 25 | 23 | 17 | 5 | 13
Participants | 25 | 23 | 17 | 5 | 13

13. Other Pre Specified Outcome: PD-1 Levels
Description: Measured at baseline and during treatment. Summarized descriptively by median, minimum, maximum and interquartile range. Overall response and complete response will be correlated with each measure using Wilcoxon rank sum test. The relationship between each measure and time to event measures will be evaluated using Cox proportional hazard models.
Time Frame: Up to 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: PD-L1 Levels
Description: as for outcome 13
Time Frame: Up to 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: PD-L2 Levels
Description: as for outcome 13
Time Frame: Up to 1 year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Markers of Immune Modulation
Description: Summarized descriptively by median, minimum, maximum, and interquartile range (continuous factors) or frequency distribution (categorical factors) at each time point. Patterns over time summarized by absolute difference or relative change. Changes across time will be assessed using paired analyses, including Wilcoxon signed rank tests for continuous measures and McNemar's tests for categorical measures. Overall response and complete response will be correlated with continuous factors using Wilcoxon rank sum tests. Jitplots will be used to visually examine differences between groups for continuous factors. Overall response and complete response will be correlated with categorical factors using Fisher's exact tests.
Time Frame: Baseline to up to 1 year
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Immune Profiles
Description: as for outcome 16
Time Frame: Baseline to up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Arm A (CLL) | Arm B (NHL) | Arm C (CLL With Richters) | Arm A (Continuation Phase) | Arm C (Continuation Phase)
All-Cause Mortality (participants affected / at risk) | 18/25 | 14/23 | 13/17 | 3/5 | 9/13
Serious Adverse Events (participants affected / at risk) | 15/25 | 9/23 | 8/17 | 3/5 | 6/13
Other Adverse Events (participants affected / at risk) | 25/25 | 22/23 | 14/17 | 5/5 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (CLL) (N=25) | Arm B (NHL) (N=23) | Arm C (CLL With Richters) (N=17) | Arm A (Continuation Phase) (N=5) | Arm C (Continuation Phase) (N=13)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 2 (3) | 2 (2) | 2 (2) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (CLL) (N=25) | Arm B (NHL) (N=23) | Arm C (CLL With Richters) (N=17) | Arm A (Continuation Phase) (N=5) | Arm C (Continuation Phase) (N=13)
Anemia (Blood and lymphatic system disorders) | 23 (69) | 17 (87) | 14 (41) | 4 (18) | 13 (52)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 8 (15) | 9 (21) | 5 (9) | 4 (6) | 6 (22)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (15) | 9 (16) | 7 (12) | 3 (5) | 2 (3)
Vomiting (Gastrointestinal disorders) | 5 (7) | 5 (6) | 5 (5) | 1 (1) | 1 (3)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 6 (7) | 4 (5) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Lymphocyte count decreased (Investigations) | 3 (4) | 6 (22) | 5 (6) | 0 (0) | 3 (3)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (34)
Neutrophil count decreased (Investigations) | 11 (20) | 7 (18) | 7 (11) | 4 (10) | 3 (7)
Platelet count decreased (Investigations) | 19 (65) | 10 (46) | 12 (32) | 5 (39) | 10 (50)
White blood cell decreased (Investigations) | 5 (8) | 10 (27) | 5 (7) | 3 (3) | 1 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (33) | 14 (28) | 9 (15) | 3 (8) | 7 (20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (23) | 8 (16) | 5 (7) | 3 (3) | 3 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (3) | 2 (4) | 4 (7) | 3 (16)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT02332980/Prot_SAP_000.pdf